CLINICAL TRIAL: NCT03751449
Title: Exercise and Nutrition Intervention in Older Breast Cancer Survivors - The WIN CA Study
Brief Title: Exercise and Nutrition Education in Improving Physical Function and Quality of Life in Older Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: i 67518; NCI-2018-01704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 67518 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Cancer Survivor; Inactivity; Obesity; Overweight; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Sedentary Behavior; Obesity; Overweight | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (active treatment) (Experimental): Participants complete a home-based aerobic and resistance exercise program and receive nutrition education for 12 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (waitlist) (Active Comparator): Participants are placed on a waitlist for 12 weeks and then complete a home-based aerobic and resistance exercise program and receive nutrition education for 12 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive nutrition education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Exercise Intervention — Complete home-based aerobic and resistance exercise program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well exercise and nutrition education work in improving physical function and quality of life in older breast cancer survivors. Exercise and nutrition education may help to improve the level of fitness, cardiovascular health, and quality of life in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of a home-based aerobic and resistance exercise and nutrition education intervention in overweight or obese, sedentary, older (65 years and above) breast cancer survivors on physical function (6-minute walk test) and quality of life compared to standard of care.

SECONDARY OBJECTIVES:

I. To assess the effect of a home-based aerobic and resistance exercise and nutrition education intervention on diet quality, sleep, anxiety, depression, source of motivation for exercise, and immune function in overweight or obese, sedentary, older (65 years and above) breast cancer survivors compared to standard of care.

EXPLORATORY OBJECTIVES:

I. To determine how body composition (dual X-ray absorptiometry [DEXA]) and weight maintenance are affected by a 12-week aerobic and resistance exercise training program among older (65 years and above), sedentary, overweight and obese breast cancer survivors.

II. To compare differences in the above outcomes among older (65 years and above), sedentary, overweight and obese breast cancer survivors who completed a home-based aerobic and resistance exercise training program versus those who did not receive the intervention, standard of care.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I (ACTIVE TREATMENT): Participants complete a home-based aerobic and resistance exercise program and receive nutrition education for 12 weeks.

GROUP II (WAITLIST): Participants are placed on a waitlist for 12 weeks and then complete a home-based aerobic and resistance exercise program and receive nutrition education for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with a history of breast cancer who have completed treatment >=3 months ago (not including hormonal therapy, Zometa, or other non-chemotherapy/radiation cancer treatment at the discretion of the principal investigator)
* Physically inactive, defined as not meeting 150 minutes or 2 hours and 30 minutes a week of vigorous-intensity exercise
* Overweight or obese, defined as having a body mass index (BMI) between 26 kg/m^2 and 42 kg/m^2, inclusive
* Meeting criteria for participation in low to moderate risk exercise based on the American College of Sports and Medicine (ACSM) guideline
* Providing informed consent indicating understanding the investigational nature of this study by signing an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedures

Exclusion Criteria:

* Metastatic breast cancer
* Orthopedic or neuromuscular disorders that preclude participation in exercise
* Any history of myocardial infarction (MI), angina pectoris, or congestive heart failure
* High risk for moderate exercise based on ACSM risk classification
* Pregnant or nursing
* Unwilling or unable to follow protocol requirements
* Any condition which - in the investigator?s opinion - deems the participant an unsuitable candidate to participate in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Activity levels for all participants will be collected using the Fitbit applications and a weekly activity log. | Up to 2 years
  Will measure the effect on physical function (6-minute walk test). Activity levels for all participants will be collected using the Fitbit applications and/or a weekly activity log.
Quality of life as assessed by the Self Geriatric Assessment Measure (GA-Self Assessment) | Up to 2 years
  Will measure the effect of a home-based aerobic and resistance exercise and nutrition education intervention on quality of life.

SECONDARY OUTCOMES:
Diet quality as assessed by the ASA24 website | Up to 2 years
  Will measure the effect of a home-based aerobic and resistance exercise and nutrition education intervention on diet quality.
Sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Up to 2 years
  The PSQI measures the quality and pattern of sleeps in adults. There are 19 items. Each item is weighted on a 0-3 interval scale.
Anxiety and the effect of a home-based aerobic and resistance exercise and nutrition education intervention | Up to 2 years
  Will measure anxiety as assessed by the State Trait Anxiety Inventory (STAI-Y1)e STAI questionnaire consists of 40 questions with 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. The scores for each subtest range from 20 to 80, with higher scores indicating higher levels of anxiety
motivation for exercise as assessed by the Behavioral Regulation for Exercise Questionnaire (BREQ-2) | Up to 2 years
  A 19 item questionnaire that measures the stages of the self-determination continuum with respect to motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me)
Centers for Epidemiologic Studies Depression Scale (CESD-R) | Up to 2 years
  A self reported 20 item scale that measures depressive symptoms. A higher score denotes greater depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States